CLINICAL TRIAL: NCT07305025
Title: Pelvic Pain Electro-Acupuncture: Randomized Study for Symptom Liberation
Brief Title: Pelvic Pain Electro-Acupuncture
Acronym: PEARL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 910176
Record Dates: First submitted 2025-11-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Pain; Endometriosis
Keywords: pelvic pain; endometriosis; acupuncture; sexual function; quality of life; pelvic floor muscle function
MeSH Terms: conditions — Pelvic Pain; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, electroacupuncture (Experimental): Frequency: 3 sessions per week for 3 weeks. Needle retention time: ~30 minutes per session. Electroacupuncture at a frequency of 2 Hz Electroacupuncture Stimulation Parameters Electroacupuncture will be administered at a frequency of 2 Hz, as this has been shown to stimulate the release of endogenous opioids, including endorphins and enkephalins. These neuropeptides contribute to pain modulation and inflammation reduction via activation of the body's natural analgesic pathways (7). Additionally, low-frequency stimulation at 2 Hz has been associated with parasympathetic nervous system activation, which may further enhance pain relief by reducing stress-related sympathetic activity and promoting a relaxed physiological state. This dual mechanism makes 2 Hz electroacupuncture a suitable intervention for chronic and inflammatory pain conditions. Electrode placement and treatment duration will be standardized across participants to ensure consistency in stimulation intensity, needle depth
  Interventions: Device: Electro acupuncture
- Control (No Intervention): Waiting as usual prior to surgery

INTERVENTIONS:
Device: Electro acupuncture — Frequency: 3 sessions per week for 3 weeks. Needle retention time: ~30 minutes per session. Electroacupuncture at a frequency of 2 Hz Electroacupuncture Stimulation Parameters Electroacupuncture will be administered at a frequency of 2 Hz, as this has been shown to stimulate the release of endogenous opioids, including endorphins and enkephalins. These neuropeptides contribute to pain modulation and inflammation reduction via activation of the body's natural analgesic pathways (7). Additionally, low-frequency stimulation at 2 Hz has been associated with parasympathetic nervous system activation, which may further enhance pain relief by reducing stress-related sympathetic activity and promoting a relaxed physiological state. This dual mechanism makes 2 Hz electroacupuncture a suitable intervention for chronic and inflammatory pain conditions. Electrode placement and treatment duration will be standardized across participants to ensure consistency in stimulation intensity, needle depth
  Arms: Intervention, electroacupuncture

SUMMARY:
The aim of the study is to investigate if a series of up to 9 treatment sessions of electroacupuncture can be used to alleviate pain in women with suspected endometriosis, scheduled for diagnostic laparoscopy

DETAILED DESCRIPTION:
1. Introduction

   Background:

   Endometriosis is a chronic inflammatory condition associated with significant pelvic pain, often requiring medical intervention. Globally, it is estimated that approximately 10 percent of reproductive-age females have endometriosis (1). Up to 70% of adolescent and adult females presenting for evaluation of chronic pelvic pain are diagnosed with endometriosis. While surgery and hormonal therapy are standard treatments, they may not be suitable or readily available for all patients. In addition, surgery is expensive and carries risk of complications.

   A systematic review and meta-analysis from 2023 including 331 women from six studies showed that acupuncture reduced overall pelvic pain and menstrual pain, but the evidence was low to moderate (2). The studies were non homogeneous regarding acupuncture style (Traditional Chinese, Japanese, ear acupuncture or unspecified), number of needles and duration of treatment. Another review from 2024 included 11 studies from China and three from other countries using different acupuncture techniques (3). They conclude that acupuncture is effective in alleviating dysmenorrhea and pelvic pain but the current evidence is limited and research focusing on subtypes of acupuncture is needed (3).

   Electro-acupuncture (EA) has been suggested as a promising approach to modulating pain perception and reducing inflammation. By influencing endogenous opioid release, regulating inflammatory cytokines, and improving pelvic blood flow, EA may provide effective symptom relief (4, 5). EA was more effective than conventional acupuncture in treating endometriosis related pain in a few studies (3, 6).

   Most previous studies are from China, and feasibility studies regarding type of acupuncture, duration of treatment, how women tolerate intervention and results on pelvic pain in a European setting are needed. Given the need for additional management options, particularly for women awaiting surgery or seeking alternatives to hormonal treatments, EA could offer valuable support in symptom relief.

   Aim:

   Primary aim: To assess the effect of acupuncture on pelvic pain in women with suspected endometriosis.

   Secondary aims: To assess the effect of acupuncture on pelvic floor muscle function, sexual function, quality of life.

   To determine feasibility for a larger-scale study.
2. Study Design Type: Randomized Controlled Trial, Pilot study, non-blinded. Sample Size: 36 women with suspected endometriosis randomized to either acupuncture treatment or standard care. Women in the acupuncture group (n=18) will receive treatment in separate 3-week periods/blocks.

   Duration: Three weeks of acupuncture treatment with follow-up at end of treatment and 2-3 months post-treatment (day of surgery).
3. Inclusion & Exclusion Criteria

   Inclusion Criteria:

   Women aged 18-45 years referred for diagnostic laparoscopy with suspicion of endometriosis Experiencing moderate to severe pelvic pain Willing to commit to the treatment schedule and follow-up Understanding Norwegian or English to be able to communicate and fill out questionnaires

   Exclusion Criteria:

   Pregnancy Use of opioid pain relief Concurrent participation in other pain management trials.
4. Intervention

   Rationale for point selection:

   Traditional Chinese Medicine (TCM) approaches treatment based on pattern differentiation, where diagnosis is guided by symptom presentation and observable signs. TCM recognizes multiple patterns for conditions like endometriosis, typically six distinct patterns. A key concept in TCM related to endometriosis is "qi and blood stagnation," a term that describes symptoms such as distension or sharp pain. While all cases of endometriosis in TCM include aspects of this pattern, the underlying TCM causes may vary. This protocol is designed to address the clinical presentation associated with qi and blood stagnation, making it standardized and broadly applicable across different cases.

   Electro-Acupuncture Treatment:

   Frequency: 3 sessions per week for 3 weeks. Needle retention time: ~30 minutes per session. Electroacupuncture at a frequency of 2 Hz Electroacupuncture Stimulation Parameters Electroacupuncture will be administered at a frequency of 2 Hz, as this has been shown to stimulate the release of endogenous opioids, including endorphins and enkephalins. These neuropeptides contribute to pain modulation and inflammation reduction via activation of the body's natural analgesic pathways (7). Additionally, low-frequency stimulation at 2 Hz has been associated with parasympathetic nervous system activation, which may further enhance pain relief by reducing stress-related sympathetic activity and promoting a relaxed physiological state. This dual mechanism makes 2 Hz electroacupuncture a suitable intervention for chronic and inflammatory pain conditions.

   Electrode placement and treatment duration will be standardized across participants to ensure consistency in stimulation intensity, needle depth, and session frequency. Acupuncture is dose-dependent, its effectiveness is influenced by treatment frequency and duration. It is thought more frequent sessions help reinforce therapeutic effects, particularly for chronic conditions. Treating pelvic pain from suspected endometriosis three times per week for three weeks ensures consistent stimulation of acupuncture points, for a sustained effect.

   Standardized point description

   KI-14 (Sì Mǎn) Location: 2 cun below the umbilicus and 0.5 cun lateral to the midline Needle Angle: Perpendicular insertion 0.5 to 1 cun Depth: Avoid deep needling to prevent penetrating peritoneal cavity in thin patients

   ST-28 (Shuidao) Location: 3 cun inferior to the umbilicus and 2 cun lateral to the midline, in the lower abdomen.

   Needle Angle: Perpendicular. Depth: 0.5-1.5 cun. Caution: Avoid deep needling to prevent injury to the peritoneal cavity in thin patients.

   LI 4 (Hegu) Location: On the dorsum of the hand, between the first and second metacarpal bones, at the midpoint of the second metacarpal bone, close to its radial border.

   Needle Angle: Perpendicular or oblique proximally toward the wrist. Depth: 0.5-1.0 cun. Contraindicated in pregnancy.

   Liv 3 (Tai Chong) Location: On the dorsum of the foot, in the depression distal to the junction of the first and second metatarsal bones.

   Needle Angle: Perpendicular or slightly oblique toward the first metatarsal space.

   Depth: 0.5-1.5 cun.

   Sp 6 (Sanyinjiao) Location: 3 cun superior to the prominence of the medial malleolus, on the posterior border of the tibia.

   Needle Angle: Perpendicular or oblique proximally. Depth: 0.5-1.5 cun. Contraindicated in pregnancy

   Sp 8 (Diji) Location: 3 cun inferior to Sp 9, on the line connecting Sp 9 and the medial malleolus, on the posterior border of the tibia.

   Needle Angle: Perpendicular. Depth: 0.5-1.5 cun. SP-10 (Xuehai) Location: On the medial aspect of the thigh, 2 cun superior to the superior border of the patella, in the bulge of the vastus medialis muscle.

   Needle Angle: Perpendicular. Depth: 0.5-1.5 cun.

   Traditional Considerations of Acupuncture Point Protocol SP6 (Sanyinjiao) - Regulates the uterus, calms pain SP8 (Diji) - for acute dysmenorrhea LV3 (Taichong) - Moves Liver Qi, reduces stagnation-related pain. Commonly used for menstrual pain, and stress relief.

   SP-10 (Xuehai) Regulates Menstruation,for menstrual disorders related to blood deficiency or stasis.

   Ki14 (Sì Mǎn) Moves Qi and Blood, alleviating pain, Irregular menstruation, dysmenorrhea ST-28 (Shuidao) - Regulates Menstruation & the Uterus, Common in gynecological treatments.

   LI4 (Hegu) is known for its strong analgesic (pain-relieving) effects and is often used for headaches, facial pain, and general pain syndromes.

   Acupuncture Needles This study will use Scarborough CJ100 acupuncture needles (0.25mm gauge, 25mm length). These needles are made from surgical-grade stainless steel (SUS304) with a coiled copper handle and loop, traditional to Chinese acupuncture. They are silicone-coated for smooth insertion and come with a guide tube for precise placement.

   ES-130 Electroacupuncture Unit - Waveform and Current ES-130 electroacupuncture unit uses an asymmetric bi-phasic pulse waveform with a phase duration of 100µs. For this study, a 2Hz current will be applied, selected from the unit's adjustable frequency range of 0-500Hz. This specific frequency is chosen for its effect on endorphin release and pain modulation (5, 8).
5. Outcome Measures

   Primary Outcomes:

   Changes in pain intensity measured via validated pain scale NRS (9, 10). Strongest, weakest, average pain last week + actual pain, all NRS scale 0 - 10 Pain catastrophizing scale (11) Type of pain (12) Amsterdam complex pelvic pain scale (13) Changes in quality of life (QoL) using a standardized questionnaire SF-36 (14). Change in pain medication use

   Secondary Outcomes:

   Changes in sexual function (FSFI, FSDS-r)(15) Pelvic ultrasound findings as an objective measure of muscle contractility (16) Changes in levator hiatal area at rest and contraction. Changes in levator hiatal anteroposterior diameter. Other outcomes from World endometriosis research foundation questionnaire

   User experience:

   How did the women experience participation in trial? What do they suggest could be done differently in future larger scale study?
6. Data Collection & Analysis

   Pre-treatment baseline assessment:

   Questionnaires Ultrasound Post-treatment assessment: At the end of the 3-week acupuncture period Questionnaires Follow-up assessments: At 2-3 months post-treatment (day of surgery) Questionnaires Ultrasound Result of surgery: confirmation of endometriosis at surgery according to revised American Fertility Society Score and histologically or other explanation to pain (adherances etc)
7. Statistics Descriptive statistics for background variables Changes in outcomes over time: Mixed models Changes in outcomes at day of surgery between intervention and control group: t-test and Mann-Whitney U-test
8. Power analyses We used this web page for power analyses: Power/Sample Size Calculator We assume that women have NRS 8 at inclusion and that women receiving acupuncture have a reduction to NRS 5 at day of surgery (SD 3). With a power and 0.8 and p-value 0.05, we would need 16 women in each group. We assume that we lose to follow up some participants, and will need to recruit 36 women, 18 in each group.
9. Risks and benefits, Clinical relevance Acupuncture is a low risk treatment method, with minimal risk of adverse events (skin infection at insertion site, mild pain) It is time consuming to fill in the questionnaire and meet for treatment Potential benefit for each woman is pain relief

Clinical relevance Surgery is expensive and medication has side effects If EA turns out to be effective as pain relief for women with chronic pelvic pain, this may benefit future patents.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years referred for diagnostic laparoscopy with suspicion of endometriosis
* Experiencing moderate to severe pelvic pain
* Willing to commit to the treatment schedule and follow-up
* Understanding Norwegian or English to be able to communicate and fill out questionnaires

Exclusion Criteria:

* Pregnancy
* Use of opioid pain relief
* Concurrent participation in other pain management trials

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 38 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
NRS | Baseline, after three months, and the day of surgery, average 6 months after baseline
  Changes in pain intensity measured via validated pain scale NRS
Quality of life SF-36 | Baseline, after three months, and the day of surgery, average 6 months after baseline
  standardized questionnaire measuring quality of life (SF-36)
Change in pain medication use | Baseline, after three months, and the day of surgery, average 6 months after baseline
  Change in pain medication use
Amsterdam complex pelvic pain scale | Baseline, after three months, and the day of surgery, average 6 months after baseline
  Changes in Amsterdam complex pelvic pain scale

SECONDARY OUTCOMES:
FSFI | Baseline, after three months, and the day of surgery, average 6 months after baseline
  Changes in sexual function FSFI
FSDS-r | Baseline, after three months, and the day of surgery, average 6 months after baseline
  Changes in sexual function (FSDS-r)
levator hiatal dimensions | Baseline and the day of surgery, average 6 months after baseline
  Chenges in levator hiatal area and anteroposterior diameter measured at rest and contraction

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Volløyhaug, PhD, Principal Investigator — St.Olavs Hopsital

IPD SHARING:
Plan to Share IPD: No
few participants included. It might be possibel to identify study participants based on characteristica such as day of surgery, age, BMI

REFERENCES:
- See also: Related Info — https://www.stolav.no/kliniske-studier/effekt-av-elektroakupunktur-pa-bekkensmerte-hos-kvinner-med-underlivssmerter-eller-endometriose/